CLINICAL TRIAL: NCT02905864
Title: Effect of Liraglutide on Body Weight and Pain in Overweight or Obese Patients With Knee Osteoarthritis: A Randomised, Double Blind, Placebo-controlled, Parallel Group, Single-centre Trial
Brief Title: Liraglutide 3 mg for Knee Osteoarthritis
Acronym: LOSEIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henrik Gudbergsen (Other)
Collaborators: Novo Nordisk A/S (Industry); Cambridge Weight Plan Limited (Industry)
Responsible Party: Sponsor-Investigator, Henrik Gudbergsen, MD, PhD, Parker Research Institute
Organization: Parker Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 137.00
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis; Obesity
Keywords: Liraglutide; Liraglutide 3 mg; Osteoarthritis; Obesity
MeSH Terms: conditions — Osteoarthritis; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide 3 mg (Experimental): Arm description: Subjects will be up titrated to liraglutide 3 mg QD and stay on that dose for the remainder of the 52-week drug intervention period.
  Drug: Liraglutide 3 mg QD administered in a 6 mg/mL, 3 mL pen for subcutaneous injection.
  Dose escalation scheme: Initial dosage of 0.6 mg per day, escalated bi-weekly by 0.6 mg to 3 mg per day over a total of 8 weeks.
  Interventions: Drug: Liraglutide 3 mg (Saxenda)
- Liraglutide 3 mg placebo (Placebo Comparator): Arm description: Subjects will be up titrated to liraglutide 3 mg placebo QD and stay on that dose for the remainder of the 52-week drug intervention period.
  Drug: Liraglutide 3 mg placebo QD administered in a 6 mg/mL drug equivalent volumes, 3 mL pen for subcutaneous injection.
  Dose escalation scheme: Initial dosage of a 0.6 mg drug equivalent volume per day, escalated bi-weekly by an 0.6 mg drug equivalent volume per day to a 3 mg drug equivalent volume per day over a total of 8 weeks.
  Interventions: Drug: Liraglutide 3 mg placebo

INTERVENTIONS:
Drug: Liraglutide 3 mg (Saxenda)
  Arms: Liraglutide 3 mg
Drug: Liraglutide 3 mg placebo
  Arms: Liraglutide 3 mg placebo

SUMMARY:
A randomised, double blind, placebo-controlled, parallel group, and single-centre trial investigating the effect of liraglutide on body weight and pain in overweight or obese patients with knee osteoarthritis.

Patients will be subjected to a run-in diet intervention phase (week -8 to 0) including a low-calorie diet and dietetic counselling. At week 0 patients will be randomised to receive either liraglutide 3 mg or liraglutide 3 mg placebo as an add-on to dietetic guidance on re-introducing regular foods and a focus on continued motivation to engage in a healthy lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Clinical diagnosis of knee OA (American College of Rheumatology (ACR) criteria) confirmed by radiology but restricted to definite radiographic OA at early to moderate-stages (Kellgren-Lawrence grades 1, 2, or 3)
* Age ≥ 18 years and < 75 years
* Body mass index (BMI) ≥ 27 kg/m2
* Stable body weight during the previous 3 months (< 5 kg self-reported weight change)
* Motivated for weight loss

Exclusion Criteria:

* On-going participation, or participation within the last 3 months, in an organised weight loss programme (or within the last 3 months)
* Current or history of treatment with medications that may cause significant weight gain for at least 3 months before this trial
* Current use or use within three months before this trial of GLP-1 receptor agonist, pramlintide, sibutramine, orlistat, zonisamide, topiramate, or phentermine
* Type 1 diabetes
* Type 2 diabetes treated with glucose-lowering drugs other than metformin
* Alloplasty in target knee joint (see section 6.3)
* End stage disease in target knee joint (Kellgren-Lawrence grade 4)
* Immuno-inflammatory disease
* Chronic wide-spread pain
* Pregnancy or insufficient anti-conception therapy for female fertile patients
* Breast-feeding
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x above upper normal range (UNR)
* Surgery scheduled for the trial duration period, except for minor surgical procedures
* Surgical procedures such as arthroscopy or injections into a knee within 3 months prior to enrolment
* Previous surgical treatment for obesity (excluding liposuction >1 year before trial entry)
* Thyroid stimulating hormone (TSH) outside of the range of 0.4-6.0 mIU/L
* Obesity secondary to endocrinologic or eating disorders or to treatment with medicinal products that may cause weight gain
* Family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2
* Inflammatory bowel disease
* Congestive heart failure, New York Heart Association (NYHA) class III-IV
* Diabetic gastroparesis
* History of or current diagnosis of pancreatitis (acute and/or chronic) or pancreatic cancer
* History of cancer with the exception of in-situ malignancies of the skin or cervix uteri
* History of major depressive disorder, a PHQ-9 (Patient Health Questionnaire-9) score of more than 15, or a history of other severe psychiatric disorders or diagnosis of an eating disorder
* Subjects with a lifetime history of a suicide attempt or history of any suicidal behaviour within the past month before entry into the trial
* Inability to speak Danish fluently
* A mental state impeding compliance with the program
* Use of opioids or similar strong analgesics
* Allergic reactions to the active ingredients of Saxenda, such as hypotension, palpitations, dyspnoea and oedema

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Week 0 to 52
  One of two co-primary outcomes
KOOS pain subscale | Week 0 to 52
  Two of two co-primary outcomes. The Knee injury and Osteoarthritis Outcome Score (KOOS); the pain subscale (9 items)

SECONDARY OUTCOMES:
KOOS symptom subscale | Week 0 to 52
  Knee injury and Osteoarthritis Outcome Score (KOOS); the symptoms subscale (7 items)
KOOS ADL subscale | Week 0 to 52
  Knee injury and Osteoarthritis Outcome Score (KOOS); the Activities of Daily Living (ADL) subscale (17 items)
KOOS sport and recreation subscale | Week 0 to 52
  Knee injury and Osteoarthritis Outcome Score (KOOS); the sport and recreation subscale (5 items)
KOOS health related QoL subscale | Week 0 to 52
  Knee injury and Osteoarthritis Outcome Score (KOOS); the health related quality of life (QoL) subscale (4 items)
Change in total score in the ICOAP questionnaire | Week 0 to 52
  The Intermittent and Constant Osteoarthritis Pain questionnaire (ICOAP); 11 items
Change in the constant pain subscale in the ICOAP questionnaire | Week 0 to 52
  The Intermittent and Constant Osteoarthritis Pain questionnaire (ICOAP); 5 items
Change in the intermittent pain subscale in the ICOAP questionnaire | Week 0 to 52
  The Intermittent and Constant Osteoarthritis Pain questionnaire (ICOAP); 6 items
Change in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain subscale | Week 0 to 52
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain subscale; 5 items
Change in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) stiffness subscale | Week 0 to 52
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) stiffness subscale; 2 items
Change in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) physical function subscale | Week 0 to 52
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) physical function subscale; 17 items
Proportion of participants with ≥5% weight loss | Week 0 to 52
  The proportion of patients with or with more than a 5% weight loss 52 weeks after randomization
Proportion of participants with ≥10% weight loss | Week 0 to 52
  The proportion of patients with or with more than a 10% weight loss 52 weeks after randomization
Change in BMI | Week 0 to 52
  Change in body mass index 52 weeks after randomization
Change in waist circumference | Week 0 to 52
  Change in waist circumference 52 weeks after randomization
Change in waist/hip circumference ratio | Week 0 to 52
  Change in the ratio waist circumference/hip circumference 52 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Henrik R Gudbergsen, MD, PhD, Principal Investigator — The Parker Institute
Locations (1):
- Department of Rheumatology, Frederiksberg, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poulsen AS, Stisen ZR, Skougaard M, Christensen R, Overgaard A, Gudbergsen H, Jacobsen S, Balslev-Clausen AP, Henriksen M, Kristensen LE, Bliddal H. Effect of weight loss and liraglutide on neutrophil gelatinase-associated lipocalin levels among individuals with overweight and knee osteoarthritis: Exploratory analyses of a randomized controlled trial. Osteoarthr Cartil Open. 2025 Jan 3;7(1):100562. doi: 10.1016/j.ocarto.2024.100562. eCollection 2025 Mar. PMID 39877802
- [Derived] Gudbergsen H, Overgaard A, Henriksen M, Waehrens EE, Bliddal H, Christensen R, Nielsen SM, Boesen M, Knop FK, Astrup A, Rasmussen MU, Bartholdy C, Daugaard CL, Ellegaard K, Heitmann BL, Bartels EM, Danneskiold-Samsoe B, Kristensen LE. Liraglutide after diet-induced weight loss for pain and weight control in knee osteoarthritis: a randomized controlled trial. Am J Clin Nutr. 2021 Feb 2;113(2):314-323. doi: 10.1093/ajcn/nqaa328. PMID 33471039
- [Derived] Daugaard CL, Henriksen M, Riis RGC, Bandak E, Nybing JD, Hangaard S, Bliddal H, Boesen M. The impact of a significant weight loss on inflammation assessed on DCE-MRI and static MRI in knee osteoarthritis: a prospective cohort study. Osteoarthritis Cartilage. 2020 Jun;28(6):766-773. doi: 10.1016/j.joca.2020.02.837. Epub 2020 Mar 10. PMID 32165240
- [Derived] Gudbergsen H, Henriksen M, Waehrens EE, Overgaard A, Bliddal H, Christensen R, Boesen MP, Knop FKK, Astrup A, Rasmussen MU, Bartholdy C, Daugaard C, Bartels EM, Ellegaard K, Heitmann BL, Kristensen LE. Effect of liraglutide on body weight and pain in patients with overweight and knee osteoarthritis: protocol for a randomised, double-blind, placebo-controlled, parallel-group, single-centre trial. BMJ Open. 2019 May 5;9(5):e024065. doi: 10.1136/bmjopen-2018-024065. PMID 31061017